CLINICAL TRIAL: NCT07052708
Title: Impact of Medication Adherence on Cardiovascular Outcomes in Individuals With Type 2 Diabetes and Disabilities: Nationwide Cohort Study
Brief Title: The Impact of Medication Adherence in Patients With Type 2 Diabetes and Disabilities
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Ki Hong Choi, Professor, Samsung Medical Center
Other Study IDs: MedicationAdherence_Disability
Record Dates: First submitted 2025-06-28; First posted 2025-07-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Disabilities; Type 2 Diabetes
Keywords: medication adherence
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disability: Individuals were classified as having a disability if they were officially registered as of the index date. Physical disability included conditions such as limb impairment, brain lesion, visual or auditory impairment, speech impairment, facial disfigurement, and epilepsy. Mental disability included intellectual disability, autism spectrum disorder, and psychiatric disorders.
  Interventions: Behavioral: No adherence group; Behavioral: Adherence group
- No disability: Individuals who were not officially registered with any physical or mental disability as of the index date.

INTERVENTIONS:
Behavioral: No adherence group — Patients with poor adherence was defined as medication possession ratio(MPR) <50%.
  Groups: Disability
Behavioral: Adherence group — Patients with good adherence was defined as medication possession ratio(MPR) ≥50%.
  Groups: Disability

SUMMARY:
Individuals with disabilities and type 2 diabetes tend to have worse clinical outcomes. To identify modifiable factors that may improve these outcomes, the investigators evaluated the role of medication adherence. A retrospective, cohort study was conducted using data from the Korean National Health Insurance Service (K-NHIS) database.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a well-established risk factor for cardiovascular disease (CVD). In recent years, self-care has become a central component of diabetes management, with growing emphasis on medication adherence, physical activity, and lifestyle modifications to reduce CVD risk and improve long-term outcomes. As a result, limited capacity for self-care has been increasingly recognized as a major contributor to health disparities.

Approximately 25% of individuals with disabilities have T2DM, and those with physical or mental impairments often face substantial barriers to effective self-management. These challenges-including limited mobility and reduced access to health information-can lead to poor glycemic control and heightened cardiovascular risk.

However, most prior studies have primarily focused on describing the elevated risk of CVD in individuals with disabilities. Whether suboptimal medication adherence mediates the association between disability and cardiovascular outcomes remains unclear.

Therefore, this study aims to compare medication adherence between patients with and without disabilities and to assess whether differences in adherence contribute to disparities in the incidence of CVD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who newly diagnosed T2DM between between January 1, 2010, and December 31, 2023

Exclusion Criteria:

* individuals with a history of MI, stroke, percutaneous coronary intervention, peripheral arterial disease, chronic kidney disease, or cancer before the diagnosis of diabetes were excluded.
* individuals with who already had diabetics related complication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients newly diagnosed with T2DM and without prior major cardiovascular or malignant conditions.
Sampling Method: Non-Probability Sample
Enrollment: 365295 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 10 years after diagnosed T2DM
  Composite of MI, ischemic stroke, hemorrhagic stroke, and all-cause mortality

SECONDARY OUTCOMES:
Diabetic neuropathy | 10 years after diagnosed T2DM
  Nerve damage resulting from DM
Diabetic foot without amputation | 10 years after diagnosed T2DM
  Diabetic foot complications, such as ulcers, infections, or gangrene, without any lower-extremity amputation
Diabetic foot with amputation | 10 years after diagnosed T2DM
  Diabetic foot complications who have undergone lower-limb amputation
Proliferative diabetic retinopathy | 10 years after diagnosed T2DM
  Advanced stage of diabetic retinopathy, marked by the formation of new blood vessels (neovascularization) on the retina or optic disc, which can lead to vitreous hemorrhage, tractional retinal detachment, and vision loss.
Non-proliferative diabetic retinopathy | 10 years after diagnosed T2DM
  Early stage of diabetic retinal disease, characterized by microaneurysms, intraretinal hemorrhages, and hard exudates without the presence of neovascularization.

IPD SHARING:
Plan to Share IPD: Undecided